CLINICAL TRIAL: NCT04252872
Title: A Randomized, Open-label, Oral Single Dose, Two-way Crossover Clinical Trial to Compare the Pharmacokinetics and Safety/Tolerability After Administration of HCP1401 and Co-administration of HCP0605 and HGP1405 in Healthy Male Volunteers
Brief Title: Pharmacokinetics of HCP1401 and Co-administration of HCP0605, HGP1405 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-ALCH-102
Record Dates: First submitted 2016-02-23; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A (Experimental): Period 1 : HCP0605+HGP1405
  Period 2 : HCP1401
  Interventions: Drug: HCP0605; Drug: HGP1405; Drug: HCP1401
- Sequence B (Experimental): Period 1 : HCP1401
  Period 2 : HCP0605+HGP1405
  Interventions: Drug: HCP0605; Drug: HGP1405; Drug: HCP1401

INTERVENTIONS:
Drug: HCP0605
Drug: HGP1405
Drug: HCP1401

SUMMARY:
A randomized, open-label, oral single dose, two-way crossover clinical trial to compare the pharmacokinetics and safety/tolerability after administration of HCP1401 and co-administration of HCP0605 and HGP1405 in healthy male volunteers

DETAILED DESCRIPTION:
The purpose of this study is to investigate the pharmacokinetics and safety/tolerability after administration of HCP1401 and co-administration of HCP0605, HGP1405 in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteer, age 19~45 years
2. Weight is not less than 55kg, no more than 90kg and Body Mass Index(BMI) is not less than 18 kg/m2 , no more than 27 kg/m2
3. Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in kidney, liver, cardiovascular system, respiratory system, endocrine system, or neuropsychiatric system.
2. Subjects who judged ineligible by the investigator.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
AUClast | pre-dose(0h), 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 22, 48, 72, 96, 120, 144 h post-dose
  Area under the plasma concentration versus time curve
Cmax | pre-dose(0h), 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 22, 48, 72, 96, 120, 144 h post-dose
  Peak Plasma Concentration

SECONDARY OUTCOMES:
AUCinf | pre-dose(0h), 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 22, 48, 72, 96, 120, 144 h post-dose
Tmax | pre-dose(0h), 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 22, 48, 72, 96, 120, 144 h post-dose
T1/2 | pre-dose(0h), 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 22, 48, 72, 96, 120, 144 h post-dose
Cl/F | pre-dose(0h), 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 22, 48, 72, 96, 120, 144 h post-dose
Vz/F | pre-dose(0h), 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 22, 48, 72, 96, 120, 144 h post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea